CLINICAL TRIAL: NCT07229014
Title: Effects of a Collagen Supplement on Quality of Life, Appetite and Glycaemic Control: a Randomised, Double-blinded, Placebo-controlled, Crossover Trial in Overweight and Obese Adults.
Brief Title: Effects of a Collagen Supplement on Quality of Life, Appetite and Glycaemic Control
Acronym: GluCol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Rousselot BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GluCol Study
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Quality of Life; Appetite; Sleep; Mood; Energy; Blood Glucose Profile
Keywords: collagen; glucose; appetite; statiety; mood; sleep

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen peptide then placebo (Experimental): 2 x 5g of hydrolysed collagen peptide daily for 8 days then crossing over to the placebo
  Interventions: Dietary Supplement: Collagen peptide supplement; Other: Placebo
- Placebo then collagen peptide (Experimental): 2 x 5g of maltodextrin daily for 8 days then crossing over to the collagen peptide
  Interventions: Dietary Supplement: Collagen peptide supplement; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Collagen peptide supplement — 5 g of hydrolysed collagen peptide of bovine origin in powdered form. Taken twice daily for 8 days total.
Other: Placebo — 5 g of maltodextrin in powdered form. Taken twice daily for 8 days total.

SUMMARY:
This is a clinical trial aimed to investigate if a collagen supplement can improve quality of life, appetite and blood sugar in overweight and obese adults aged 18-65.

Hypothesis: Consumption of a collagen supplement for 8 days will improve quality of life and improve glycaemic control in comparison with a placebo in individuals overweight or with obesity with a perceived low quality of life.

Participants will be asked to:

1. Consume a collagen peptide supplement for a total of 8 days at a time
2. Fill in questionnaires about quality of life, appetite, mood and energy
3. Wear continuous glucose monitors

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy (as assessed by medical history) male or female adult, aged 18-65 years and overweight or obese (BMI 25 - 40 kg/m2).
2. Subject has an impaired quality of life, as determined by scoring at least a total of 9 on the following questions:

   1. In the past 4 weeks, did you feel you had a lot of energy? All of the time (1), most of the time (2), a good bit of the time (3), some of the time (4), a little of the time (5), and none of the time (6) (number 27 from SF-36 questionnaire) Version 3.0 [01/10/2025] Page 11 of 20
   2. In the past 4 weeks, have you felt calm and peaceful? All of the time (1), most of the time (2), a good bit of the time (3), some of the time (4), a little of the time (5), and none of the time (6) (number 26 from SF-36 questionnaire)
   3. In the past 2 weeks, did you have any difficulties with sleeping? Not at all (1), small amounts (2), moderate amounts (3), a great deal (4), an extreme amount (5), all the time (6) (number 3 from WHOQoL-100)
3. Participant has an email address, internet access, a compatible smartphone and is willing and able to maintain internet access throughout the trial to complete virtual visits via video conference and to engage with mobile apps to answer electronic questionnaires.
4. Subject is willing and able to comply with all study procedures, including consumption of the supplement daily, CGM use for 22 days total (2 x 11 days), complete standardised meal tests, and fill out health questionnaires.
5. Subject is willing to take a supplement of bovine animal origin.
6. Openness to participate in an online interview at the end of the study.

Exclusion Criteria:

1. Participant has a history or presence of uncontrolled and/or clinically important pulmonary, cardiac, hepatic, renal, endocrine (including type 1 and 2 diabetes), hematologic, immunologic, neurologic (e.g., Alzheimer's or Parkinson's diseases), psychiatric (including unstable depression and/or anxiety disorders) or biliary disorders.
2. Participant has a clinically important gastrointestinal (GI) condition that would potentially interfere with the evaluation of the study product [e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation, severe constipation (in the opinion of the investigator), history of frequent diarrhoea, history of surgery for weight loss, gastroparesis, systemic disease that might affect gut motility according to the investigator, medication managed reflux and/or clinically important lactose intolerance.
3. Participant has a history of chronic insomnia (defined as insomnia at least 3 d/week over the past month), a diagnosed sleep disorder (e.g., OSA), or a chronic medical condition that may impact energy/fatigue levels, in the judgment of the investigator.
4. Participant is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded.
5. Participant has a known allergy, intolerance, or sensitivity to any of the ingredients in the study product, including bovine animal products.
6. Participant has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
7. Participant has experienced any major trauma or any other surgical event within three months of Virtual Visit 1.
8. Participant has unstable use of a medication or supplement that the investigator considers may affect the outcomes of the trial.
9. Participant is currently in another biomedical research study or has been in the 30 days before screening.
10. Participant is an employee of, or has a financial interest in Darling Ingredients Inc.
11. The individual has a condition the investigator believes would interfere with his ability to provide informed consent and to comply with the study protocol, which might confound the interpretation of the study results, or put the participant at undue risk.
12. Participant is a vegan or vegetarian or excludes bovine products for cultural or religious reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life scores | Baseline and 8 days
  Quality of life (QoL) scores based on the composite scoring of the 36-item Short Form Survey (SF-36)

SECONDARY OUTCOMES:
Postprandial appetite, hunger, fullness, satiety or desire to eat | 15, 30, 60, 120 and 180 minutes post-meal
  Postprandial appetite (hunger, fullness, satiety or desire to eat), energy and mood after consumption of a standardised challenge meal, measured using a digital visual analogue scale (VAS)
Mood | Baseline and 7 days
  Mood measured using the Positive and Negative Affect Schedule Short Form (PANAS-SF) for positive affects (PA), negative affects (NA) and affect balance scores.
Energy and fatigue | Baseline and 7 days
  Energy and fatigue measured using the Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) for fatigue, energy and overall scores
Sleep | Baseline and 8 days
  Sleep measured with the Pittsburgh Sleep Quality Index (PSQI) for Global PSQI score and component scores of sleep quality, latency, duration, efficiency, disturbances and daytime dysfunction.
Glycaemic variability | From baseline to 8 days
  Glycaemic variability, including overall mean blood glucose, fasting blood glucose, daytime mean blood glucose, daytime glucose variability (CV), % time within range and number of hypoglycaemic events, measured via a continuous glucose monitor (CGM)
Postprandial glucose response | Continous monitoring up to 5 hours post-meal
  Postprandial glucose response to a standardised breakfast expressed in difference in glucose Cmax, glucose Cmin, glucose Tmax, glucose Tmin and area under the curve, measured using continuous glucose monitor (CGM)
Habitual diet | Baseline only
  Habitual diet assessed via the European Prospective Investigation into Cancer and Nutrition (EPIC) food frequency questionnaire (FFQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolic Research Unit (KCL, Waterloo Campus), London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No